CLINICAL TRIAL: NCT06402630
Title: A Phase 2 Double-blind, Multicentre, Placebo Controlled, Parallel Group Design to Assess the Efficacy, Safety and Dose Response Characterisation of STS01 for the Treatment of Mild-moderate Alopecia Areata (AA)
Brief Title: A Phase 2 Placebo Controlled, Clinical Trial Designed to Assess the Efficacy, Safety and Dose Response Characterisation of STS01 for the Treatment of Mild-moderate Alopecia Areata (AA)
Acronym: SOT01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soterios Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOT01; 2021-004145-20 (EudraCT Number)
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Alopecia Areata
Keywords: alopecia areata; alopecia; areata; aa; autoimmune; hair loss; hair; autoimmune hair; follicle
MeSH Terms: conditions — Alopecia Areata; Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.25% Dose (Experimental): Once daily, STS-01 topical cream applied to affected area of the head
  Interventions: Drug: STS01
- 0.5% Dose (Experimental): Once daily, STS-01 topical cream applied to affected area of the head
  Interventions: Drug: STS01
- 1% Dose (Experimental): Once daily, STS-01 topical cream applied to affected area of the head
  Interventions: Drug: STS01
- 2% Dose (Experimental): Once daily, STS-01 topical cream applied to affected area of the head
  Interventions: Drug: STS01
- Placebo (Placebo Comparator): Once daily, topical cream applied to affected area of the head (without API)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STS01 — Participants are block randomised to be treated with 0.25%, 0.5%, 1.0%, 2% STS-01 or a matching placebo control topically once daily for 6 months with a 2-month follow up.
  Arms: 0.25% Dose; 0.5% Dose; 1% Dose; 2% Dose
Drug: Placebo — Participants are block randomised to be treated with 0.25%, 0.5%, 1.0%, 2% STS-01 or a matching placebo control topically once daily for 6 months with a 2-month follow up.
  Arms: Placebo

SUMMARY:
A Phase 2 double-blind, multi-site, placebo-controlled, parallel-group design to assess the efficacy, safety and dose-response characterisation of STS-01 for the treatment of mild- moderate alopecia areata.

DETAILED DESCRIPTION:
STS-01 is being developed to address the need for an effective, safe and convenient non-steroidal topical treatment for mild-moderate alopecia areata. The product builds on a mechanism with a well-established safety profile in dermatology, and existing evidence of its effectiveness in this condition through targeting key relevant cytokines. STS-01 has been modified to maximise the effectiveness of this mechanism and offer a cosmetically elegant topical cream. The study aims to assess the effectiveness, safety and dose-response characteristics of STS-01 for the treatment of mild-moderate alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

1. Active alopecia areata (less than 50% SALT score, present for at least 6 months)
2. Not currently receiving treatment for hair loss
3. Eighteen years of age or more
4. Affected skin with normal appearance and no grossly evident epidermal alteration such as scaling or follicular abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in Alopecia areata severity measured using the Severity of Alopecia Tool (SALT) at 6 months | 6 Months
  Alopecia areata severity measured using the Severity of Alopecia Tool (SALT) at 6 months. Targeting patients with <50 SALT (less than 50% hair loss).

SECONDARY OUTCOMES:
Regrowth area measured by graphical measuring of the size of the patch | 6 months
  Regrowth area measured by graphical measuring of the size of the patch
Global assessment using the Clinical Global Impression (CGI) score | 6 Months
  Global assessment using the Clinical Global Impression (CGI) score
AA quality of life measured using Subject Alopecia Areata Symptom Impact Scale (AASIS) | 6 Months
  AA quality of life measured using Subject Alopecia Areata Symptom Impact Scale (AASIS)
AA quality of life measured using Alopecia Areata Quality of Life Index (AAQLI) 0-25 | 6 months
  AA quality of life measured using Alopecia Areata Quality of Life Index (AAQLI) 0-25

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Queen Margaret Hospital, Glasgow, Dunfirmline
  - St Lukes Hospital, Bradford, Little Horton Lane
  - Royal Alexandra Children's Hospital, Brighton
  - University Hospital Coventry & Warwickshire, Coventry
  - Queen Elizabeth University Hospital, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Queen Anne Street Medical Centre Limited, London
  - Norfolk and Norwich University Hospital, Norwich
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No